CLINICAL TRIAL: NCT01259934
Title: Nordic Randomized Phase III Trial of Two Different Durations of Adjuvant Therapy With Intermediate-dose Interferon Alfa-2b in Patients With High-risk Melanoma
Brief Title: Nordic Adjuvant IFN Melanoma Trial
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Johan Hansson, PI, Department of Oncology-Pathology, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Nordic-IFN-melanoma trial
Record Dates: First submitted 2010-12-10; First posted 2010-12-14 (Estimated); Last update posted 2010-12-14 (Estimated); Status verified 2010-12

CONDITIONS: Melanoma; Adjuvant Therapy
Keywords: Randomized Phase III trial; Adjuvant therapy; Interferon; Melanoma
MeSH Terms: conditions — Melanoma | interventions — Interferon-alpha2b; Introns

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Arm A (No Intervention): Observation only - no therapy
- Arm B Interferon 1 year (Experimental): Interferon Therapy: Induction: IFN-alfa2b, 10 MU (flat dose), SC, 5 days/week, 4 weeks Maintenance: IFN-alfa2b, 10 MU (flat dose), 3 days/week, SC, 12 months
  Interventions: Drug: Interferon-alpha2b - 1 year
- Arm C Interferon 2 years (Experimental): "Two year arm" Induction: IFN-alfa2b, 10 MU (flat dose), SC, 5 days/week, 4 weeks Maintenance: IFN-alfa2b, 10 MU (flat dose), 3 days/week, SC, 24 months
  Interventions: Drug: Interferon-alpha2b - 2 years

INTERVENTIONS:
Drug: Interferon-alpha2b - 1 year — Induction: IFN-alpha2b, 10 MU (flat dose), SC, 5 days/week, 4 weeks Maintenance: IFN-alpha2b, 10 MU (flat dose), 3 days/week, SC, 12 months
  Other Names: Intron-A
  Arms: Arm B Interferon 1 year
Drug: Interferon-alpha2b - 2 years — Induction: IFN-alfa2b, 10 MU (flat dose), SC, 5 days/week, 4 weeks Maintenance: IFN-alfa2b, 10 MU (flat dose), 3 days/week, SC, 24 months
  Other Names: Intron-A
  Arms: Arm C Interferon 2 years

SUMMARY:
The aim of this study is to evaluate the effect of giving adjuvant treatment with intermediate doses of interferon-alpha2b to patients operated for high risk melanoma. Patients are randomly assigned to either observation only or interferon treatment for 2 different durations. The outcome with respect to overall survival, relapse-free survival, side effects and quality of life is analysed.

DETAILED DESCRIPTION:
This is an open multicenter, prospective randomised phase III trial evaluating the efficacy of two different schedules of Interferon-alpha2b (IFN-alpha2b) administered in an adjuvant setting after adequate surgery in high risk cutaneous melanoma patients (T4N0M0/TxN1-2M0). The patients have been operated for either a thick primary melanoma (> 4 mm) without evidence of distant metastasis or have undergone surgery for regional lymph node metastases.

The study consists of a control arm (A) and two treatment arms, B and C. The outcome in arms B and C with adjuvant treatment with IFN-alpha2b will be compared to the outcome of arm A in which the patients will only be observed after the surgery. The primary endpoint is overall survival. Secondary endpoints are relapse-free survival, safety-toxicity and health-related quality of life.

ELIGIBILITY:
Inclusion Criteria:

* T4 N0 M0 - Thick primary melanoma: > 4.0 mm Breslow depth, without lymph node involvement, or
* Tx N1-2 M0 Primary melanoma of any thickness with regional lymph node metastases confirmed by lymphadenectomy, or
* Tx N1-2 M0 Recurrent melanoma in regional lymph node(s) confirmed by lymphadenectomy.
* ECOG performance status of 0-1
* No active medical or psychiatric disorder requiring therapy that would prevent completion of protocol
* Written informed consent

Exclusion Criteria:

* Patients with unknown primary site of melanoma or primary melanoma originating apart from the skin, except subungual melanoma
* Patients who have clinical, radiological/laboratory or pathological evidence of incompletely resected melanoma or distant metastatic disease
* Patients who have had prior adjuvant radiotherapy, chemotherapy, immunotherapy including preoperative infusion or perfusion therapy
* Female patients who are pregnant or lactating

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 855 (Actual)
Dates: Start 1996-11; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
Overall survival | Evaluated at regular intervals: every 3 months for 2 years, every 6 months up to 5 years and yearly up to 10 years following randomization. Actual median follow-up is 72.4 months
  All registered deaths, not only melanoma-specific.

SECONDARY OUTCOMES:
Relapse free survival | Evaluated at regular intervals
  Time from randomization to date of first reported melanoma recurrence or death
Safety-toxicity | Regular evaluations
  All toxicities and SAEs are recorded and classified according to CTC v2.0 criteria
Health related quality of life | Regular evaluations
  Recorded by using the EORTC QLQ-C30 questionnaire at nine time points during treatment and follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Johan Hansson, MD,PhD, Study Chair — Karolinska Institutet; Steinar Aamdal, MD. PhD, Principal Investigator — Oslo University Hospital, Oslo, Norway; Lars Bastholt, MD,PhD, Principal Investigator — Odense University Hospital; Micaela Hernberg, MD, PhD, Principal Investigator — Helsinki University Central Hospital, Helsinki, Finland; Ulrika Stierner, MD PhD, Principal Investigator — Sahlgrenska University Hospital; Hans von der Maase, MD PhD, Principal Investigator — Copenhagen University Hospital, Copenhagen, Denmark
Locations (1):
- Karolinska Institutet, Karolinska University Hospital,, Stockholm, Sweden

REFERENCES:
- [Background] Bouwhuis MG, Suciu S, Collette S, Aamdal S, Kruit WH, Bastholt L, Stierner U, Sales F, Patel P, Punt CJ, Hernberg M, Spatz A, ten Hagen TL, Hansson J, Eggermont AM; EORTC Melanoma Group and the Nordic Melanoma Group. Autoimmune antibodies and recurrence-free interval in melanoma patients treated with adjuvant interferon. J Natl Cancer Inst. 2009 Jun 16;101(12):869-77. doi: 10.1093/jnci/djp132. Epub 2009 Jun 9. PMID 19509353
- [Derived] Prasmickaite L, Berge G, Bettum IJ, Aamdal S, Hansson J, Bastholt L, Oijordsbakken M, Boye K, Maelandsmo GM. Evaluation of serum osteopontin level and gene polymorphism as biomarkers: analyses from the Nordic Adjuvant Interferon alpha Melanoma trial. Cancer Immunol Immunother. 2015 Jun;64(6):769-76. doi: 10.1007/s00262-015-1686-4. Epub 2015 Apr 2. PMID 25832001
- [Derived] Hansson J, Aamdal S, Bastholt L, Brandberg Y, Hernberg M, Nilsson B, Stierner U, von der Maase H; Nordic Melanoma Cooperative Group. Two different durations of adjuvant therapy with intermediate-dose interferon alfa-2b in patients with high-risk melanoma (Nordic IFN trial): a randomised phase 3 trial. Lancet Oncol. 2011 Feb;12(2):144-52. doi: 10.1016/S1470-2045(10)70288-6. Epub 2011 Jan 20. PMID 21256809